CLINICAL TRIAL: NCT03473106
Title: Effect of the Use of Tourniquet in the Thigh: a Biomechanical Analysis on the Muscular Function of the Quadriceps in the Postoperative Period.
Brief Title: Effect of Tourniquet Use on Muscle Thigh Function.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Daniela Bravo Advis, Assistant Professor, Department of Anesthesia, University of Chile
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: OAIC 919/17
Record Dates: First submitted 2018-03-11; First posted 2018-03-22 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Pneumatic Tourniquet; Muscle Weakness
Keywords: Pneumatic Tourniquet; Postoperative Muscle Dysfunction
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Surgical side can not be randomized. Only data assessor will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical Side (Experimental): Surgical side requiring the use of a pneumatic tourniquet.
  Interventions: Device: Pneumatic tourniquet use
- Non Surgical Side (No Intervention): Contralateral side (Control Thigh).

INTERVENTIONS:
Device: Pneumatic tourniquet use — Surgery requiring a pneumatic tourniquet on the thigh
  Arms: Surgical Side

SUMMARY:
The use of a pneumatic tourniquet with the purpose of maintaining an operative field free of blood is a common practice in orthopedic surgery. Its use is associated with local and systemic consequences related to hemodynamic and reperfusion ischemia phenomena. Although is known that its use is not an innocuous measure, there is still certain degree blurriness regarding the potential metabolic and functional consequences that may result in the involved limb.

In this trial, the investigators are setting out to discriminate the effect of the pneumatic tourniquet on thigh muscle function (strength, tone and activation). The hypothesis is that the pneumatic tourniquet by itself causes a significant postoperative muscular dysfunction of the quadriceps and, thus, the main outcome will be the presence of postoperative quadriceps muscle dysfunction, defined as a fall greater than or equal to 10% of the maximal voluntary isometric contraction measured at 24 hours post surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing forefoot surgery that requires the use of a pneumatic tourniquet
* American Society of Anesthesiologists classification 1-3

Exclusion Criteria:

* Ambulatory surgery
* Adults who are unable to give their own consent
* Pre-existing neuropathy or myopathy
* Contraindication of tourniquet use
* Bilateral surgery
* Pregnancy
* Hip, thigh, knee, leg or ankle pathologies that prevent or contraindicate using a dynamometer, tonometer or surface electromyographer
* Arterial hypertension with systolic pressures above 200mmHg
* Renal failure
* Hepatic failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-04-24 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Postoperative muscle dysfunction | 24 hours
  Fall greater or equal than 10% of the voluntary isometric muscle contraction from basal

SECONDARY OUTCOMES:
Basal upper and lower extremity blood pressures | Up to 2 hours pre spinal anesthesia
  Pre spinal anesthesia measured blood pressures
Upper and lower extremity blood pressures after spinal anesthesia | 10 minutes after spinal anesthesia
  Post spinal anesthesia measured blood pressures
Arterial occlusion pressure | 10 minutes after spinal anesthesia
  Doppler estimation of arterial occlusion pressure of the lower extremity surgical side
Pneumatic tourniquet inflation pressure | 3 hours from tourniquet inflation
  Arterial occlusion pressure plus a safety margin
Pneumatic tourniquet inflation time | 3 hours from tourniquet inflation
  Time from inflation to release of the pneumatic tourniquet
Quadriceps electromyographic activation profile | 24 hours
  Basal and 24 hours (post surgery) quadriceps activation on surgical side
Quadriceps muscle tone | 24 hours
  Basal and 24 hours (post surgery) measurement of quadriceps muscle tone on surgical side
Thigh perimeter | 24 hours
  Basal and 24 hours (post surgery) bilateral measurement of thigh perimeter
Thigh pain | 24 hours
  Basal and 24 hours (post surgery) bilateral thigh pain measured with a numerical rating scale (0-10)
Postoperative measurements time | 24 hours
  Time from pneumatic tourniquet release to postoperative muscle function measurements

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universidad de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Halladin NL, Zahle FV, Rosenberg J, Gogenur I. Interventions to reduce tourniquet-related ischaemic damage in orthopaedic surgery: a qualitative systematic review of randomised trials. Anaesthesia. 2014 Sep;69(9):1033-50. doi: 10.1111/anae.12664. Epub 2014 May 7. PMID 24800642
- [Result] Estebe JP, Davies JM, Richebe P. The pneumatic tourniquet: mechanical, ischaemia-reperfusion and systemic effects. Eur J Anaesthesiol. 2011 Jun;28(6):404-11. doi: 10.1097/EJA.0b013e328346d5a9. PMID 21502865
- [Result] Horlocker TT, Hebl JR, Gali B, Jankowski CJ, Burkle CM, Berry DJ, Zepeda FA, Stevens SR, Schroeder DR. Anesthetic, patient, and surgical risk factors for neurologic complications after prolonged total tourniquet time during total knee arthroplasty. Anesth Analg. 2006 Mar;102(3):950-5. doi: 10.1213/01.ane.0000194875.05587.7e. PMID 16492857
- [Result] Tai TW, Lin CJ, Jou IM, Chang CW, Lai KA, Yang CY. Tourniquet use in total knee arthroplasty: a meta-analysis. Knee Surg Sports Traumatol Arthrosc. 2011 Jul;19(7):1121-30. doi: 10.1007/s00167-010-1342-7. Epub 2010 Dec 15. PMID 21161177
- [Result] Kam PC, Kavanagh R, Yoong FF. The arterial tourniquet: pathophysiological consequences and anaesthetic implications. Anaesthesia. 2001 Jun;56(6):534-45. doi: 10.1046/j.1365-2044.2001.01982.x. PMID 11412159
- [Result] Tuncali B, Boya H, Kayhan Z, Arac S, Camurdan MA. Clinical utilization of arterial occlusion pressure estimation method in lower limb surgery: effectiveness of tourniquet pressures. Acta Orthop Traumatol Turc. 2016;50(2):171-7. doi: 10.3944/AOTT.2015.15.0175. PMID 26969952
- [Result] Guler O, Mahirogullari M, Isyar M, Piskin A, Yalcin S, Mutlu S, Sahin B. Comparison of quadriceps muscle volume after unilateral total knee arthroplasty with and without tourniquet use. Knee Surg Sports Traumatol Arthrosc. 2016 Aug;24(8):2595-605. doi: 10.1007/s00167-015-3872-5. Epub 2015 Nov 21. PMID 26590567
- [Result] Dennis DA, Kittelson AJ, Yang CC, Miner TM, Kim RH, Stevens-Lapsley JE. Does Tourniquet Use in TKA Affect Recovery of Lower Extremity Strength and Function? A Randomized Trial. Clin Orthop Relat Res. 2016 Jan;474(1):69-77. doi: 10.1007/s11999-015-4393-8. PMID 26100254
- [Result] Kruse H, Christensen KP, Moller AM, Gogenur I. Tourniquet use during ankle surgery leads to increased postoperative opioid use. J Clin Anesth. 2015 Aug;27(5):380-4. doi: 10.1016/j.jclinane.2015.03.034. Epub 2015 May 12. PMID 25979462
- [Result] Smith TO, Hing CB. The efficacy of the tourniquet in foot and ankle surgery? A systematic review and meta-analysis. Foot Ankle Surg. 2010 Mar;16(1):3-8. doi: 10.1016/j.fas.2009.03.006. Epub 2009 May 27. PMID 20152747
- [Result] Nicholas SJ, Tyler TF, McHugh MP, Gleim GW. The effect on leg strength of tourniquet use during anterior cruciate ligament reconstruction: A prospective randomized study. Arthroscopy. 2001 Jul;17(6):603-7. doi: 10.1053/jars.2001.24854. PMID 11447547